CLINICAL TRIAL: NCT01882257
Title: Home-Based Diagnosis and Management of Sleep-Related Breathing Disorders in Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Robert G. Sitrin, M.D., Professor of Internal Medicine, University of Michigan
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM00051504; W81XWH-11-1-0826 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2013-06-17; First posted 2013-06-20 (Estimated); Results first posted 2017-01-04 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Obstructive Sleep Apnea; Hypercapnia; Spinal Cord Injury
Keywords: obstructive sleep apnea; sleep-disordered breathing; hypercapnia; spinal cord injury
MeSH Terms: conditions — Sleep Apnea, Obstructive; Hypercapnia; Spinal Cord Injuries; Sleep Apnea Syndromes | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Normal sleep breathing (No Intervention): Home-based sleep studies indicate no obstructive sleep apnea or nocturnal hypoventilation. No intervention.
- BiPAP -Auto for sleep apnea (Experimental): Patients whose home-based sleep study detects obstructive sleep apnea, but no nocturnal hypoventilation. Noninvasive ventilatory support will be prescribed according to standard clinical criteria.
  Interventions: Device: BiPAP
- BiPAP (AVAPS) for nocturnal hypoventilation (Experimental): Patients whose home-based sleep study detects nocturnal hypoventilation in the presence or absence of obstructive sleep apnea. Noninvasive ventilatory support will be prescribed according to standard clinical criteria. BiPAP/AVAPS (Phillips Respironics) is worn with a mask interface of the subject's choice. It is specifically designed to treat nocturnal hypoventilation.
  Interventions: Device: BiPAP/AVAPS (Phillips Respironics)

INTERVENTIONS:
Device: BiPAP — BiPAP-auto (Phillips Respironics)is a noninvasive positive pressure ventilation device worn with a mask interface of the subject's choice. It is used to treat obstructive sleep apnea.
  Other Names: BiPAP-auto (Phillips Respironics)
  Arms: BiPAP -Auto for sleep apnea
Device: BiPAP/AVAPS (Phillips Respironics) — BiPAP/AVAPS (Phillips Respironics) is a noninvasive positive pressure ventilation device worn with a mask interface of the subject's choice. It is specifically designed to treat nocturnal hypoventilation due to an underlying neuromuscular disorder.
  Arms: BiPAP (AVAPS) for nocturnal hypoventilation

SUMMARY:
* Patients with spinal cord injury (SCI) usually breathe without any mechanical assistance, but significant breathing problems occur often during sleep, either because the upper airway closes (obstructive sleep apnea; OSA), or because of weakness/paralysis of the breathing muscles. These problems often go unrecognized, as SCI patients face logistical barriers that cause them to refuse appropriate testing in sleep laboratories. We have devised a strategy for diagnosing sleep-disordered breathing in the patient's home, using placement of noninvasive devices that monitor breathing overnight. This project is designed to test the feasibility and utility of this strategy.
* After collecting baseline data on symptoms and medical events for four months, the home-based studies are performed noninvasively with FDA-approved devices: a type III sleep system and a recording oxygen saturation/ transcutaneous carbon dioxide monitor. If these studies identify sleep-disordered breathing, noninvasive ventilatory support is prescribed according to standard clinical practice. Over the following twelve months, the subjects monitor their symptoms daily, and answer quality-of-life questionnaires every three months. After 3, 6, and 12 months, blood tests are performed to measure blood sugar and cholesterol/lipids. Data is downloaded from the ventilator device to monitor compliance and ventilator performance. This study is designed to determine the prevalence of sleep-disordered breathing in SCI, the feasibility of home-based testing to establish the diagnosis, and the short term effects on symptoms, quality-of-life, and associated conditions (glucose intolerance, blood lipid disorders).

DETAILED DESCRIPTION:
Eligible subjects will sign informed consent, followed by:

a 4 month period of maintaining a daily log of symptoms and medical events (such as hospitalization, starting antibiotics).

An overnight sleep study will be performed in the subject's home Based on the results of the sleep study, noninvasive ventilation (BiPAP) will be prescribed, according to standard medical practice. A clinical assessment, pulmonary function tests, and blood tests (blood glucose, hemoglobin A1C, and blood lipid profile) will be performed at the same time.

Quality of life surveys will be performed at months 0, 3, 6, and 12. The daily symptom logs will be continued for 12 months. Data from the BiPAP units will be downloaded and repeat overnight monitoring to measure blood oxygen and carbon dioxide levels will be performed periodically for 12 months after BiPAP is started.

Subjects without sleep-disordered breathing will have the same clinical assessments and blood tests as subjects for whom BiPAP has been described.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* C1-T6 spinal cord injury for at least 3 months
* living within 100 miles of Ann Arbor, Michigan, USA

Exclusion Criteria:

* unable to provide informed consent
* comorbid condition that limits life expectancy to less than 1 year
* ventilator-dependent
* established diagnosis of sleep-disordered breathing
* prior use of noninvasive positive pressure ventilation (CPAP or BiPAP) for any reason (temporary suse of noninvasive ventilation during a hospitalization is permissible if it was discontinued more than 3 months prior to enrollment)
* active duty military personnel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2011-10; Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert G Sitrin, Md, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Bauman KA, Kurili A, Schotland HM, Rodriguez GM, Chiodo AE, Sitrin RG. Simplified Approach to Diagnosing Sleep-Disordered Breathing and Nocturnal Hypercapnia in Individuals With Spinal Cord Injury. Arch Phys Med Rehabil. 2016 Mar;97(3):363-71. doi: 10.1016/j.apmr.2015.07.026. Epub 2015 Aug 20. PMID 26297810

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 93 subjects were enrolled in the study. 2 subjects were found to be ineligible due to level of spinal cord injury. 91 patients remained in the study and were asked to keep daily logs of symptoms. 17 subjects were unable or unwilling to come to the first study visit.
Period: Study Origination to Beginning Therapy
Arm/Group | Normal Sleep Breathing | BiPAP -Auto for Sleep Apnea | BiPAP (AVAPS) for Nocturnal Hypoventilation
Started | 11 | 40 | 23
Started Therapy Using Device | 11 | 38 (Of the 40 who were given the device, 2 chose not to begin the actual therapy) | 22 (Of the 23 who were given the device, 1 chose not to begin the actual therapy)
Completed (Month 0 Visit Attended) | 11 | 38 | 22
Not Completed | 0 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 2 | 1
Period: Therapy Portion of Study (12 Months)
Arm/Group | Normal Sleep Breathing | BiPAP -Auto for Sleep Apnea | BiPAP (AVAPS) for Nocturnal Hypoventilation
Started | 11 | 38 | 22
Completed (Completed Study, Month 12 Final Visit) | 11 | 27 | 18
Not Completed | 0 | 11 | 4
Not completed — Withdrawal by Subject | 0 | 11 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Sleep Breathing | BiPAP -Auto for Sleep Apnea | BiPAP (AVAPS) for Nocturnal Hypoventilation | Total
Number analyzed (Participants) | 11 | 40 | 23 | 74
Age, Customized [Number; unit: participants]
  18 to 75 years | 11 | 40 | 23 | 74
Gender [Count of Participants; unit: Participants]
  Female | 2 | 5 | 3 | 10
  Male | 9 | 35 | 20 | 64
Region of Enrollment [Number; unit: participants]
  United States | 11 | 40 | 23 | 74

OUTCOME MEASURES:

1. Primary Outcome: Prevalence of Sleep-disordered Breathing in Spinal Cord-injured Adults
Description: After enrollment, the subject completes symptom logs for four months to collect baseline data. At that point, the home-based sleep study is performed, and the results determine whether the subject has sleep-disordered breathing. The primary outcome to be measured in this study is to determine the prevalence and type of sleep-disordered breathing in subjects with spinal cord injury. These results in turn determine the type of positive pressure device to be prescribed, as detailed in the description of the study arms. Therefore, the arm distribution is itself a primary outcome of this study.
Time Frame: Month 4 after enrollment
Measure: Number; unit: participants
Groups:
- Entire Tested Population: All groups are considered together because this outcome is simply identifying what portion of the defined population (People with Spinal Cord Injury) have which types of sleep disordered breathing
Arm/Group | Entire Tested Population
Number analyzed (Participants) | 74
participants
  Sleep disordered breathing without hypercapnia | 40
  Sleep-disordered breathing with hypercapnia | 23
  Normal sleep breathing | 11

2. Primary Outcome: The Frequency of Technical Errors Related to the Home-based Overnight Testing.
Description: All testing was done overnight, and if the home-based overnight test was inadequate, that portion of the testing was repeated (also overnight).
Time Frame: Overnight testing (4-13 hours)
Measure: Number; unit: participants
Groups:
- Entire Tested Population: All groups are considered together because in determining the efficiency and reliability of home-based overnight testing, there is no difference between the three groups
Arm/Group | Entire Tested Population
Number analyzed (Participants) | 74
participants
  HSAT (Home Sleep Apnea Test) | 6
  Transcutaneous pCO2/SpO2 Monitor | 9

3. Other Pre Specified Outcome: Short Term Effects on Daily Symptoms and Medical Events
Description: The subjects keep daily logs of certain symptoms and events (pulmonary symptoms that require escalated care, pulmonary infections, doctor visits, hospitalizations, antibiotic use, symptoms of unstable blood pressure). These data are collected throughout the study period
Time Frame: Months 0-16 after enrollment
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Short Term Effects of Noninvasive Ventilatory Support on Quality of Life
Description: At month 4 of the study, and every 3 months therafter for 12 months, the subjects will complete standardized questionnaires on quality of life, focusing on general well being, mood, pain, and sleepiness.
Time Frame: Months 4-16
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Short Term Effects of Noninvasive Ventilatory Support on Glucose and Lipid Metabolism
Description: When home-based sleep testing is performed, and at 3, 6, and 12 months afterward, subjects will have blood tests to determine if treatment of sleep-disordered breathing has any effects on glucose intolerance/diabetes and/or blood cholesterol/lipid levels
Time Frame: Months 4-16
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Identify Clinical Features That Are Predict or Are Associated With the Severity of Sleep-disordered Breathing
Description: Clinical features (neck and waist circumference, body mass index, level and duration of spinal cord injury, lung function tests, questionnaire results) will be analyzed to determine if certain attributes predict the presence or severity of sleep-disordered breathing.
Time Frame: Month 4 after enrollment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 months from the allocation to the device (or not) to the end of the study
Arm/Group | Normal Sleep Breathing | BiPAP -Auto for Sleep Apnea | BiPAP (AVAPS) for Nocturnal Hypoventilation
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/40 | 0/23
Other Adverse Events (participants affected / at risk) | 0/11 | 0/40 | 0/23

LIMITATIONS AND CAVEATS:
Although this study demonstrates that home-based overnight testing can identify sleep-disordered breathing in patients with spinal cord injury, it remains an individual clinical decision whether facility-based testing is preferable for some.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes